CLINICAL TRIAL: NCT05255172
Title: Physiological Mechanisms Affecting Exercise Capacity in Patients With Heart Failure - an Exercise Intervention Study Evaluated With Several Modalities
Brief Title: Exercise Intervention in Patients With Heart Failure With Preserved and Reduced Ejection Fraction
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-05044
Record Dates: First submitted 2022-01-20; First posted 2022-02-24 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure New York Heart Association (NYHA) Class II; Heart Failure New York Heart Association (NYHA) Class III

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised exercise (Experimental): The exercise intervention will include 2 supervised sessions of ergometer cycling with a warm up period of 10 minutes and 20 minutes of cycling at the aerobic intensity below the anaerobic threshold as determined from baseline results. Patients in the exercise arm will have 1 unsupervised exercise session where the participants walk or bicycle for 30 minutes at an intensity experienced as somewhat hard (Borg 13) according to the Borg Rating of Perceived Exertion Scale.
  Interventions: Other: Supervised Exercise
- Standard of Care (No Intervention): The control group will receive advise to continue to live as usual. After 4 and 8 weeks, participants in the control group will be contacted by telephone for inquiry of general wellbeing. No other interventions will be performed in the control group.

INTERVENTIONS:
Other: Supervised Exercise — 12 weeks of supervised aerobic exercise individually adapted to exercise capacity according to a VO2 peak test
  Arms: Supervised exercise

SUMMARY:
The objective of this study is to assess by what physiological mechanisms patients with heart failure benefit from exercise. Effects of an exercise intervention will be assessed for both central (heart and lungs) and peripheral (muscle fiber and mitochondria) factors.

DETAILED DESCRIPTION:
A randomized, non-blinded prospective intervention trial. Patients randomized to exercise intervention will undergo supervised aerobic training on ergometer cycle for 12 weeks whilst control group receives standard care. Before and after the intervention, all participants will undergo cardiac magnetic resonance imaging (cardiac MR) examinations, Ventilation/Perfusion Single Photon Emission Computed Tomography (V/P SPECT), Cardiopulmonary exercise tests, muscle biopsies and blood sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Signs and symptoms of heart failure
2. Age ≥50 years
3. Stable chronic heart failure (no hospitalizations within past month, no new medications past month)
4. Able to understand and follow exercise prescription
5. Currently physically inactive (less than 150 minutes/week moderate intensity exercise)

Exclusion criteria:

1. Currently or within the past 6 months been involved in cardiac rehab with exercise
2. Devices or implants not compatible with magnetic resonance imaging or exercise testing
3. Any orthopedic or medical condition affecting participation in testing and training
4. Signs of acute ischemia during baseline cardiopulmonary exercise testing
5. Participation in other clinical trials that may affect results
6. Moderate or severe valvular disease
7. Atrial fibrillation
8. Moderate or severe chronic obstructive pulmonary disease
9. NYHA class IV

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen uptake (VO2peak) | 12 weeks intervention
  a change in maximal oxygen uptake (VO2 peak) of 2 ml/min/kg

SECONDARY OUTCOMES:
Health related quality of life | 12 weeks intervention
  Change in Health related quality of life assessed with Kansas City Cardiomyopathy Questionnaire (KCCQ). KCCQ scores are scaled from 0 to 100 and summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Cardiac volumes and function | 12 weeks intervention
  Change in cardiac volumes and function assessed using Cardiac MR indicating effects of the exercise intervention as compared to the control group
Perfusion gradients on Ventilation / Perfusion Single Photon Emission Computed Tomography (V/P SPECT) | 12 weeks intervention
  Change in pulmonary congestion quantified by V/P SPECT
Mitochondrial function | 12 weeks intervention
  Change in mitochondrial number and function using respirometry indicating effects of the exercise intervention as compared to the control group

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University Hospital Lund, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No